CLINICAL TRIAL: NCT06763627
Title: The Effectiveness of Gamification-Based Learning Versus Traditional Classroom Teaching in Acute Cholecystitis and Pancreatitis Education Among Medical Students: A Quasi-Experimental Study
Brief Title: The Effectiveness of Gamification vs. Traditional Teaching in Undergraduate Medical Education
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IR.IUMS.REC.1403.896
Record Dates: First submitted 2025-01-03; First posted 2025-01-08 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Medical Education; Gamification
Keywords: Gamification; Boardgame; Medical Education; Medical Student; General Surgery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Gamification group (Experimental): The gamification group will consist of teams of three to four members, who will engage in the board game under the supervision of the supervising investigator for one hour.
  Interventions: Other: Gamification ( Board game )
- Class group (Active Comparator): The class group will consist of individuals who will attend a one-hour traditional, lecture-based session led by a faculty member in general surgery
  Interventions: Other: Traditional lecture-based teaching

INTERVENTIONS:
Other: Gamification ( Board game ) — A three- or four-player board game will be designed to teach acute cholecystitis and pancreatitis. The game has two stages: educational (houses 1-9) and reinforcement (houses 10-30). Players roll dice and move their pieces to answer various questions such as multiple-choice, true/false, matching, puzzles, and scenario-based problem-solving. Each player starts with three hearts, and if they land on one of the three red "trap" spaces and answer incorrectly, they lose one heart. Yellow spaces introduce random events like gaining or losing hearts. One space features a general knowledge question for variety. Players must achieve a point threshold in the educational section to move to the reinforcement section, and the highest scorer at the end of the hour wins. Groups of 3 or 4 students will play for one hour under the supervision of the investigator.
  Arms: Gamification group
Other: Traditional lecture-based teaching — Students will attend a standard one-hour lecture delivered by a general surgery faculty member, covering the same topics. PowerPoint presentations prepared by the research team will ensure consistency with the game content.
  Arms: Class group

SUMMARY:
This study will evaluate the effectiveness of a gamification-based learning method (board game) versus traditional teaching (lecture) in enhancing the knowledge of acute cholecystitis and pancreatitis among medical students in the general surgery ward at Rasoul Akram Hospital. This study will be conducted as an extra-curricular program, using pre- and post-tests to determine the effectiveness of gamification in general surgery learning within undergraduate medical education. The board game will incorporate innovative educational strategies to engage students in learning about acute cholecystitis and pancreatitis

ELIGIBILITY:
Inclusion Criteria:

* Medical students in their clinical externship in the general surgery ward.
* Willingness to participate voluntarily.

Exclusion Criteria:

* Previous knowledge or exposure to acute cholecystitis and pancreatitis.
* Lack of consent or inability to attend the sessions.
* Medical students not currently assigned to general surgery clinical rotations.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2025-01-15 (Actual); Primary Completion 2025-04-15 (Actual); Study Completion 2025-05-30 (Actual)

PRIMARY OUTCOMES:
Change in knowledge of acute cholecystitis and pancreatitis | Baseline (pre-intervention) and immediately after the intervention
  Change in Test Scores from Pre-test to Immediate Post-test, Containing 20 Multiple-Choice Questions and 10 Short-Answer Questions, Assessing Knowledge of Acute Cholecystitis and Pancreatitis: A Comparison Between Two Groups

SECONDARY OUTCOMES:
Retention of knowledge on acute cholecystitis and pancreatitis | 6 weeks after the intervention
  Retention of Knowledge Assessed by Test Scores 6 Weeks Post-Intervention, Containing 20 Multiple-Choice Questions and 10 Short-Answer Questions, on Acute Cholecystitis and Pancreatitis: A Comparison Between Two Groups

CONTACTS AND LOCATIONS:
Locations (1):
- Iran University of Medical Sciences, Tehran, Tehran Province, Iran